CLINICAL TRIAL: NCT03079947
Title: Effectiveness of Circulating DNA for Predicting the Relapse and Overall Survival in Non-hodgkin Lymphoma Patients
Brief Title: Effectiveness of Circulating DNA for Predicting the Relapse and Overall Survival in NHL Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-1149
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Diffuse Large B Cell Lymphoma; Peripheral T Cell Lymphoma
Keywords: Circulating DNA; Diffuse Large B Cell Lymphoma; Peripheral T-Cell Lymphoma; prognosis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating DNA from plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-hodgkin Lymphoma: 300 Non-hodgkin Lymphoma patients (age >=18y) without previous treatment would be administered, including DLBCLs and PTCLs.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of circulating DNA from peripheral blood for predicting the prognosis and relapse in DLBCL and PTCL patients.

DETAILED DESCRIPTION:
The investigators plan to prospectively involve 300 Non-hodgkin Lymphoma patients, including both diffuse large B cell lymphomas and peripheral T cell lymphomas without previous treatment from Peking Union Medical College Hospital.

The following parameters were collected: age, sex, subtype, Eastern Cooperative Oncology Group (ECOG) performance status (PS), Ann Arbor stage (I-IV), presence of B symptoms, number and type of involved sites, prognostic index including International Prognostic Index (IPI) for DLBCLand PIT for PTCL based on medical record review.

All patients would have regular treatment and follow up in PUMCH. During the follow up, treatment response was evaluated by contrast enhanced computed tomography or PET-CT.

The peripheral blood would be collected and circulating DNA would be tested at the time of diagnosis, interim of treatment, end of treatment, 1 year follow-up, 1.5 year of follow-up, 2 year of follow up, 3 year of follow-up and disease progression or relapse. TCR/BCR domain would be sequenced by high-throughput sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed diffuse large B cell lymphoma (DLBCL nos, PCNSL, ALK+ DLBCL, DLBCL/BL) or peripheral T cell lymphoma (AITL, ALCL, PTCL nos, NK/T nasal type, EATL, HSTL)
2. no treatment before
3. hCG(-)
4. 18 years old to 80 years old

Exclusion Criteria:

1. other tumors
2. severe infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed to be diffuse large B cell lymphoma or peripheral T cell lymphoma without any previous treatment in Peking Union Medical College Hospital (PUMCH) would be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
relapse of the disease | within 3 years
progression free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roschewski M, Dunleavy K, Pittaluga S, Moorhead M, Pepin F, Kong K, Shovlin M, Jaffe ES, Staudt LM, Lai C, Steinberg SM, Chen CC, Zheng J, Willis TD, Faham M, Wilson WH. Circulating tumour DNA and CT monitoring in patients with untreated diffuse large B-cell lymphoma: a correlative biomarker study. Lancet Oncol. 2015 May;16(5):541-9. doi: 10.1016/S1470-2045(15)70106-3. Epub 2015 Apr 1. PMID 25842160
- [Background] Kurtz DM, Green MR, Bratman SV, Scherer F, Liu CL, Kunder CA, Takahashi K, Glover C, Keane C, Kihira S, Visser B, Callahan J, Kong KA, Faham M, Corbelli KS, Miklos D, Advani RH, Levy R, Hicks RJ, Hertzberg M, Ohgami RS, Gandhi MK, Diehn M, Alizadeh AA. Noninvasive monitoring of diffuse large B-cell lymphoma by immunoglobulin high-throughput sequencing. Blood. 2015 Jun 11;125(24):3679-87. doi: 10.1182/blood-2015-03-635169. Epub 2015 Apr 17. PMID 25887775